CLINICAL TRIAL: NCT02245035
Title: Dairy Intake and Brain Health in Aging
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Principal Investigator, In-Young Choi, Ph.D., Associate Professor, University of Kansas Medical Center
Other Study IDs: 12884
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Aged Healthy Volunteer
Keywords: Glutathione; Dairy consumption; Brain; Humans

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low dairy intake: 1 serving/day or less of dairy food characterized at enrollment using 24 hr dietary recall
- Moderate Dairy Intake: 1-2 servings/day of dairy food characterized at enrollment using 24 hr dietary recall
- Recommended Dairy Intake: Greater than 3 servings/day of dairy food characterized at enrollment using 24 hr dietary recall

SUMMARY:
The purpose of this study is to learn if dairy food consumption may help brain health in aging by protecting nerve cells from oxidative damage.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 60-85 years of age.
2. Good general health with no concomitant diseases, which would be expected to interfere with the study
3. BMI range 20-35 kg/m2

Exclusion Criteria:

1. Presence of any central neurological disease with the potential to impair cognition(e.g., brain tumor, stroke, epilepsy, motor neuron disease, multiple sclerosis, Alzheimer disease, Parkinson's disease) or prior major head trauma with loss of consciousness
2. Presence of an active unstable and life-threatening systemic illness (e.g., cancer)
3. Presence of major psychiatric disorder within the past 3 years including depression, anxiety, and alcohol (over 3 drinks per day or total of 18 per week) or drug abuse (DSM-IV criteria; Geriatric Depression Score>6)
4. Presence of diabetes mellitus (defined as a clinical diagnosis or use of an anti-diabetic agent) and metabolic syndrome
5. Use of psychoactive and investigational medications
6. Subjects with MRI contraindications such as pacemaker, aneurysm clips, artificial heart valves, metal fragments, foreign objects or claustrophobia. All subjects subjects will receive a structural MRI as part of this study. Individuals with evidence of infection, infarction, neoplasm or other lesions will be excluded. Individuals found to have abnormalities in their structural MRI will be referred to their primary physician for further evaluation and management.
7. Pregnancy
8. Special diet regimens such as lactose free or vegan

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy elderly individuals with an age range of 60-85 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cerebral glutathione (GSH) levels measured by magnetic resonance spectroscopy (MRS) | Baseline
Dietary dairy food intake measured using 7-day diet recording | 1 week, prior to MRS scan

CONTACTS AND LOCATIONS:
Overall Officials: In-Young Choi, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States